CLINICAL TRIAL: NCT07260253
Title: Investigating the Benefits of Remotely-Supervised Neuromodulation In Primary Progressive Aphasia
Brief Title: Remotely-supervised Neuromodulation in PPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RF1AG085565 (NIH); RF1AG085565 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-12-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Primary Progressive Aphasia(PPA); Progressive Aphasia; Progressive Aphasia in Alzheimer's Disease; Logopenic Progressive Aphasia (LPA); Logopenic Variant Primary Progressive Aphasia; Logopenic Variant of Primary Progressive Aphasia (LPA)
Keywords: lvPPA; PPA; logopenic variant PPA; transcranial direct-current stimulation; tDCS; neuromodulation; speech therapy; speech-language pathology; logopenic; teletherapy; remote; virtual
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two arms: sham or active remotely-supervised transcranial direct current stimulation (RS-tDCS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Language Therapy with Active Stimulation (Experimental): Transcranial direct current stimulation (tDCS) is a type of non-invasive brain stimulation. 1.5 milliamp (mA) of current will be delivered via electrodes in saline-soaked sponges placed on the left and right sides of the head. The stimulation will be delivered for 20 minutes, 5 times weekly, in the participant's home setting while the participant engages in virtual speech-language training. Sessions are monitored by study personnel.
  Interventions: Behavioral: Lexical Retrieval Cascade Treatment; Device: Remotely Supervised Transcranial Direct Current Stimulation
- Language Therapy with Sham Stimulation (Sham Comparator): Transcranial direct current stimulation (tDCS) is a type of non-invasive brain stimulation. During sham stimulation 1.5 milliamp (mA) of current will be delivered for a brief period and then turned off. Current will be delivered via electrodes in saline-soaked sponges placed on the left and right sides of the head. Sham will be delivered for 20 minutes, 5 times weekly, in the participant's home setting while the participant engages in virtual speech-language training. Sessions are monitored by study personnel.
  Interventions: Behavioral: Lexical Retrieval Cascade Treatment; Device: Remotely Supervised Transcranial Direct Current Stimulation

INTERVENTIONS:
Behavioral: Lexical Retrieval Cascade Treatment — Participants work on producing spoken and written names of personally relevant target items using a self-cueing hierarchy. Treatment focuses on the use of strategies that capitalize on spared cognitive-linguistic abilities to support word retrieval. The participant completes two (one hour each) teletherapy sessions per week with a clinician plus 30 minutes of additional independent, computer-based practice exercises 3 times per week.
  Other Names: LRCT
Device: Remotely Supervised Transcranial Direct Current Stimulation — tDCS is a type of non-invasive brain stimulation. 1.5 milliamp (mA) of current will be delivered via electrodes in saline-soaked sponges placed on the left and right sides of the head. During sham stimulation 1.5 milliamp (mA) of current will be delivered for a brief period and then turned off. The stimulation will be delivered for 20 minutes, 5 times weekly, in the participant's home setting while the participant engages in computer-delivered speech-language training. Sessions are monitored by study personnel.

SUMMARY:
The goal of this clinical trial is to learn whether remotely-supervised transcranial direct-current stimulation (RS-tDCS) can improve speech and language treatments for individuals with logopenic variant primary progressive aphasia (lvPPA). tDCS is a form of brain stimulation where a low-level electrical current is delivered to the brain through electrodes placed on the head.

The main questions the trial aims to answer are:

* Is it feasible to do RS-tDCS with virtual speech therapy?
* How can brain magnetic resonance imaging scans (MRIs) predict how well someone will benefit from RS-tDCS with virtual speech therapy?

Researchers will compare active RS-tDCS stimulation to sham stimulation (where there is no active stimulation, but participants feel stimulation effects at the beginning and end of the session).

Participants will:

* Travel to either the University of California, San Francisco (UCSF) or the University of Texas at Austin (UT Austin) one time for in-person testing, an MRI scan, and training on how to use the RS-tDCS equipment
* Meet with a speech-language pathologist for pre-treatment testing on Zoom for 2 weeks
* Participate in speech-language therapy and independent practice on Zoom 5 days a week for 4 weeks, using either active tDCS stimulation or sham
* Complete post-treatment testing on Zoom for 1-2 weeks
* Complete follow-up testing 2 months after completion of treatment

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for primary progressive aphasia (PPA)
* Meets diagnostic criteria for logopenic variant PPA
* Score of 20 or higher on the Mini-Mental State Examination
* Adequate hearing and vision (with hearing or vision aids, if needed)
* Has a study partner that can co-enroll in the study and attend pre-treatment training as well as continue to be present for teleconference meetings, as needed
* Able and willing to undergo MRI brain scan
* Access to high speed internet and basic experience using a computer and the internet
* Individuals should be fluent speakers of English

Exclusion Criteria:

* Speech and language deficits better accounted for by another neurological disorder
* Does not meet diagnostic criteria for logopenic variant PPA
* Score of less than 20 on the Mini-Mental State Examination
* Does not have a study partner who can co-enroll in the study
* Contraindications for tDCS or MRI scan (History of seizures, head injury, craniotomy, skull surgery or fracture; History of severe or frequent migraines; Metallic implant in head or any metal in head; Pacemaker or cardioverter-defibrillator or any other stimulator; Chronic skin problems; Pregnancy)
* History of stroke, epilepsy, or significant brain injury

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in spoken naming | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change in percent correctly named trained/untrained pictures

SECONDARY OUTCOMES:
Change on Communication Confidence Rating Scale for Aphasia | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change on self-rating scale evaluating communication confidence in different settings for persons with aphasia. A higher score indicates greater confidence, with minimum and maximum values of 0 and 100.
Change on Aphasia Impact Questionnaire | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change on patient reported outcome measure for persons with aphasia; characterizes activities, participation and emotional state/wellbeing using a 5-point pictorial rating scale. A higher score indicates greater impact of aphasia, with minimum and maximum values of 0 and 84.
Theoretical Framework of Acceptability Questionnaire | one month after onset of treatment
  The Theoretical Framework of Acceptability questionnaire is a measure developed for healthcare interventions to identify characteristics of interventions that may be improved or that were well-received.
Acceptability and Perception of Change Survey | one month after onset of treatment
  The Acceptability and Perception of Change Survey characterizes perceived response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maya L Henry, PhD, Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - UCSF Memory and Aging Cener, San Francisco, California
  - University of Texas, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including behavioral and MRI/fMRI data from 80 individuals with lvPPA and limited data from study partners, will be shared via the ICPSR repository. Data will be available at publication or within 9 months of database lock, and accessible for at least 10 years. Publicly shared datasets will exclude identifiable information, audio/video files, and non-skull-stripped imaging. Additional data may be shared via IRB-approved data-sharing agreements.
Time Frame: De-identified clinical trial data (participant level and summary level data, raw and processed) will be made available at the time of publication of the primary results or within 9 months of database lock, whichever comes first. We will also include relevant datasets as supplementary material accompanying articles submitted to PubMed Central. Data will be publicly available for 10 years following the end of the award and by request thereafter.
Access Criteria: De-identified data will be accessible to researchers and the broader scientific community. Publicly available datasets will be hosted on the ICPSR repository and accessible via DOI. Additional data (e.g., voice samples) may be accessed through an IRB-approved data-sharing agreement, which will require users to commit to secure data handling and non-identification of participants.

REFERENCES:
- [Background] Dial HR, Hinshelwood HA, Grasso SM, Hubbard HI, Gorno-Tempini ML, Henry ML. Investigating the utility of teletherapy in individuals with primary progressive aphasia. Clin Interv Aging. 2019 Feb 25;14:453-471. doi: 10.2147/CIA.S178878. eCollection 2019. PMID 30880927
- [Background] Henry ML, Hubbard HI, Grasso SM, Dial HR, Beeson PM, Miller BL, Gorno-Tempini ML. Treatment for Word Retrieval in Semantic and Logopenic Variants of Primary Progressive Aphasia: Immediate and Long-Term Outcomes. J Speech Lang Hear Res. 2019 Aug 15;62(8):2723-2749. doi: 10.1044/2018_JSLHR-L-18-0144. Epub 2019 Aug 7. PMID 31390290
- See also: University of Texas Aphasia Research and Treatment Lab — https://slhs.utexas.edu/research/aphasia-research-treatment-lab